CLINICAL TRIAL: NCT04310358
Title: Online Perceptual Modules and Spaced Learning, a Modern Approach to Teaching Left Ventricular Systolic Assessment to Medical Students.
Brief Title: Online Perceptual Modules and Spaced Learning, a Modern Approach to Teaching LVEF Assessment to Medical Students.
Acronym: MAP-ETT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19.360
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Medical Education

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLM group 1 (Experimental): Participants will do a pretest (Test 1), the 4 short PLMs, an immediate post-test (Test 2) and a remote post-test (Test 1).
  Interventions: Other: 4 short PLMs group 1
- PLM group 2 (Experimental): Participants will do a pretest (Test 2), the 4 short PLMs, an immediate post-test (Test 1) and a remote post-test (Test 2).
  Interventions: Other: 4 short PLMs group 2

INTERVENTIONS:
Other: 4 short PLMs group 1 — Participants will take the 4 short PLMs on the visual estimation of LVEF. They will also take a pretest, an immediate post-test and a remote post-test at 1 month. Test 1 (pre-test), Test 2 (immediate post-test), Test 1 (remote post-test)
  Arms: PLM group 1
Other: 4 short PLMs group 2 — Participants will take the 4 short PLMs on the visual estimation of LVEF. They will also take a pretest, an immediate post-test and a remote post-test at 1 month. Test 2 (pre-test), Test 1 (immediate post-test), Test 2 (remote post-test)
  Arms: PLM group 2

SUMMARY:
This study is designed to:

1. Create 4 short PLMs aimed at improving visual estimation of LVEF on TTE images.
2. Design a study to determine if these online PLMs can be used to increase the ability of medical students to estimate LVEF on TTE images and create long term retention of this skill.

The hypothesis of the study is that several short PLM sessions over a period of approximately 1 month will improve the ability of third- and fourth-year novice medical students in echocardiography to visually estimate LVEF using TTE images.

DETAILED DESCRIPTION:
Echocardiography is increasingly used in the field of acute care for the diagnosis and monitoring of patients. However, echocardiography is a difficult tool to master and the recommendations for training in echocardiography require several tests to be performed and interpreted. In a context of growing training needs, this long process of supervised learning, even if it has been proven, presents difficulties, particularly the limited access to patients and experts.

Perceptual learning modules (PLMs) represent an alternative modality to teach image interpretation, and are already used in other fields where expertise is largely based on the ability to recognize patterns. Placed on digital platforms, PLMs offer a series of images and the learner must answer a question within a short time. Each response is followed by immediate feedback (the correct answer). Thus, the learner can learn to quickly extract the useful information, in this case, the left ventricle ejection fraction (LVEF) by viewing a large number of exams in a short period of time, and by receiving quality feedback every time.

Methods:

Perceptual learning modules (PLMs)

* PLMs will be assembled on the online platform using the image bank.
* Their objective is to improve visual estimation of LVEF.
* 96 TTE exams from the image bank will be used to build 4 distinct PLM modules of 24 images each.
* The answer key (LVEF) for each image set in the PLMs and performance tests will be created by an echocardiography trained cardiologist using visual assessment of LVEF and 3D measurements of LVEF.
* For every exam within a PLM, the 3 standard echocardiographic views (apical 4-chamber, apical 2-chamber, and apical long axis views) will be shown simultaneously and playing in a continuous loop for a maximum of 20 seconds.
* The online platform will allow the participants to enter their visual estimation of the LVEF (an integer between 0 and 100%).
* If no answer is entered after 20 seconds, the images will disappear, and the platform will force the participants to enter an answer before providing feedback
* Feedback will be displayed following each participant answer for a maximum of 10-seconds. During the feedback phase, the same three views will be shown, but they will be accompanied by the participants' answer and by the validated LVEF. Since LVEF by 3D assessment is the most accurate, it will be used as the validated answer for the PLMs.
* Each module will be composed of

  * 6 exams with a validated LVEF of less than 30%
  * 6 exams with a validated LVEF of 30-39%
  * 6 exams with a validated LVEF of 40-49%
  * 6 exams with a validated LVEF of 50% or more
* The order of the exams within a module will be determined at random by the online platform.
* The maximum duration of each module will be 12 minutes.
* Each exam will only be seen once. There will be no exam repetition within the modules or performance test.
* It will be possible to pause the module between exams. During a pause, the images will not be shown.

Performance tests 1 and 2

* Two performance tests of 20 exams each will be created using exams from the image banks distinct from the 96 used for the PLMs.
* The objective of the tests is to measure the participants' ability to accurately estimate LVEF (not to teach the skill),
* During testing, TTE exams will be presented like they are during the PLMs (same three views looping continuously, maximum of 20 seconds per exam)
* As in the PLMs, the online platform will allow the participants to enter their estimation of the LVEF as an integer between 0 and 100.
* However, after the participants' answer is entered, the platform will directly move on to the next exam and no feedback will be given (the validated LVEF will not be given).
* The maximum duration of each test will be 6 minutes and 40 seconds.

Study chronology

Each participant will be issued a unique secured login into the online platform. After providing informed consent and before beginning the study, each participant will complete a short survey on their demographic characteristics and clinical experience, checking specifically for exclusion criteria. After being given instructions on how the TTE exams are displayed on the platform, how to enter their visual estimations, and the difference between the testing and the learning portions of the project, all participants will take a 20-exam performance pretest to measure their baseline ability to visually estimate LVEF. Which version of the test they take will be determined at random by the platform (see below for randomization strategy).

Immediately after the pretest, the first PLM will be done. Then, the platform will lock itself for 5 days. Once this 5-day period has past, the platform will reopen, and the participant will be able to complete the second PLM within the next 5 days. Access to the platform will then again be blocked for another 5 days, after which the third PLM will become available, again for 5 days. Finally, 5 days later, the participants will be able to complete the fourth and final PLM. The exact PLM sequence each participant will complete will be determined at random by the platform. Upon completing the fourth and last PLM, all participants will take a 20-exam immediate post-test. Four weeks (28 days) after completing the last PLM and the immediate post-test, the remote post-test will be available for a one-week period. This test will contain the same test version taken as a pretest. Given the 43 to 65 day delay between both tests, and given the large number of TTE exams visualized by each participant during the study, it is considered unlikely that participants would be able to remember the exams from one test to another.

During the study, whenever a test or a PLM becomes available, the participants will automatically be informed by email. Any participants who fails to complete one of these steps within the allowed time will be excluded from the results analysis.

Randomization strategy

To minimize any bias in the eventuality that the level of difficulty of the two performance tests were to be different, participants will be randomized by blocks of 2 to one of two sequences of performance tests. These two sequences are:

* Test 1 (pre-test), Test 2 (immediate post-test), Test 1 (remote post-test)
* Test 2 (pre-test), Test 1 (immediate post-test), Test 2 (remote post-test)

Furthermore, participants will be randomly assigned a PLM sequence by the platform to avoid biases in the eventuality that the difficulty of the modules differed from one another.

ELIGIBILITY:
Inclusion Criteria:

* Third- or fourth-year medical students
* Access to a computer with high speed internet (no smartphone or tablet since the images would be too small)

Exclusion Criteria:

* Previous formal echocardiographic training (transthoracic, transesophageal or FOCUS echocardiography)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Impact of the spaced online 4 short PLMs on the ability to correctly visually estimate LVEF during a remote post-test (1 month). | Change between baseline (pre-test) and remote post-test (1 month)
  The mean absolute deviation of the participants' visual estimations from the validated answer (expert estimate) will be used as a measure of the precision of the estimations.

SECONDARY OUTCOMES:
Impact of the online perceptual modules on the ability to correctly estimate LVEF during an immediate post-test (module validation). | Change between baseline (pre-test) and immediately after the fourth PLM online session.
  The mean absolute deviation of the participants' visual estimations from the validated answer (expert estimate) will be used as a measure of the precision of the estimations.
The progression (improvement of performance) of the participants' ability to correctly assess LVEF throughout the completion of the 4 modules. | At the end of the fourth online session, on an average of 15 to up to 30 days.
  The evolution of the participants' accuracy in LVEF estimation during the PLMs could allow us to estimate a learning curve for our study group.
The fluency (time to answer) of each participant as they progress through the study protocol. | At baseline (pretest), immediately after the fourth PLM online session and on remote post-test (1 month).
  The mean response time in seconds to the different tests.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Mercier-Laporte, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No